CLINICAL TRIAL: NCT05597267
Title: The MIRIA Acne Scar Study
Acronym: MIRIA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: AVAVA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AV-22-002
Record Dates: First submitted 2022-10-24; First posted 2022-10-28 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Acne Scars - Mixed Atrophic and Hypertrophic
Keywords: Laser Treatment; Acne Scars; MIRIA Laser; Laser; AVAVA; All Skin Types; Scars
MeSH Terms: conditions — Hypertrophy; Cicatrix

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Treatment with the MIRIA Laser (Experimental): 3-4 experimental treatments at 4-6 week intervals
  Interventions: Device: MIRIA Laser

INTERVENTIONS:
Device: MIRIA Laser — 4-6 experimental treatments at 4-6 weeks intervals

SUMMARY:
This study is being conducted to evaluate the performance and efficacy of the AVAVA MIRIA Laser Skin System treatment on acne scars. Participants will be treated with the MIRIA laser at least 4 times with each treatment spaced 4-6 weeks apart. The improvement of acne scars will be evaluated at 1 month and 3 months with a possibility of 6 months evaluation after the fourth treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subjects 18-65 years of age
* Acne scars on the face
* Able and willing to comply with all study procedures and at home care; and,
* Able and willing to give informed consent.

Exclusion Criteria:

* Hypersensitive to light in the near infrared wavelength region
* On medication known to increase sensitivity to sunlight
* Seizure disorder triggered by light
* Takes or has taken oral isotretinoin, such as Accutane®, within the last six months
* Use of topical over the counter or prescription retinoids such as Retinol creams, gels, Tazarotene, Tretinoin, Adapalene, within the last 30 days
* Active acne or rosacea
* Active localized or systemic infection, or an open wound or abscess in area being treated
* Significant systemic inflammatory disease or illness, such as lupus, or an illness localized in area being treated
* Common acquired nevi that are predisposed to the development of malignant melanoma
* Current or prior herpes simplex in the target treatment area
* Is receiving or has received gold therapy
* Currently enrolled in an investigational drug or device trial, or has received an investigational drug or was treated with an investigational device within in the area to be treated 6 months prior to study entry
* Facial cosmetic procedures in the target areas within previous 6 months (e.g., laser or other energy-based device treatment, microdermabrasion, injection of dermal filler)
* Micro-needling and/or chemical peel on the target treatment area in the past 3 months
* Injection of cosmetic neurotoxins such as botulinum toxin in the treatment areas within the previous 3 months of standard duration toxins, and 6 months for long lasting neurotoxin therapy
* Significant uncontrolled concurrent illness, such as diabetes mellitus, hypertension, or cardiovascular disease
* History of immunosuppression/immune deficiency disorder or currently using immunosuppressive medications
* Planned weight loss of greater than five pounds
* Facial hair in the treatment areas which would prevent evaluation of the outcome measures. For men, must be clean shaven in the area of treatment
* Any condition or situation which, in the investigators opinion, may put the subject at significant risk, may confound study results or may interfere significantly with the subject's participation
* Is pregnant or of childbearing potential and not using medically effective birth control, or has been pregnant in the last 3 months, is currently breast feeding or planning a pregnancy during the study.
* Has had unprotected sun exposure within four weeks of treatment, including the use of tanning beds or plans for unprotected sun exposure during the course of the study,
* Has used tanning products, such as creams, lotions and sprays within four weeks prior to treatment.
* Coagulation disorder or currently using anti-platelet/anticoagulation medication, including use of aspirin, or fish oil supplements
* Taking medications that alter the wound-healing response or evidence of compromised wound healing
* Known history of keloid formation
* Known history of medical diseases that may cause koebnerization (the appearance of disease in another location), such as vitiligo, psoriasis or lichen planus
* History of skin cancer or suspicious lesions in treatment area
* Subject is relocating out of the zone of the study site (ie. Moving out of state or about 50+ miles away from study area)
* Subject has history or active melasma or other pigmentary disorders such as vitiligo.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2022-11-04 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
ECCA (échelle d'évaluation clinique des cicatrices d'acné) Grading | 3 months after the final treatment, Optional 6 months after final treatment
  A 1 point or greater reduction in facial acne scars severity using the Echelle d'Evaluation Clinique des Cicatrices d'Acne (ECCA) Score
  ECCA Global Score Limits: Lowest Score (0) to Highest Score (540)

SECONDARY OUTCOMES:
Blinded Evaluation of Treatment Imaging | From enrollment up to3 months after the final treatment, Optional up to 6 months after final treatment
  Panel of independent expert grader dermatologists will review randomized photo sets of pre- and post-treatment imaging and asked to identify the post-treatment image.
Physician Global Aesthetic Improvement Scale Scoring | Up to 3 months after the final treatment, Optional up to 6 months after final treatment
  Primary physician for the investigative site will review post-treatment imaging and score the improvement seen in the photos based on the below scale.
  5 - Much Improved 4 - Improved 3 - No Change 2 - Worse
  1 - Much Worse
Treatment Pain Assessment | Through study completion, an average of 12 months
  Treatment Pain will be assessed at all treatment visits on a standard Visual Analog Scale Ranging from a score of 0 (no pain) to 10 (maximum possible pain)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Enchantress Dermatology, Miami, Florida
  - AVAVA, Inc., Waltham, Massachusetts
  - Laser and Skin Surgery Center of New York, New York, New York

IPD SHARING:
Plan to Share IPD: No
Data is not currently being planned for sharing.